CLINICAL TRIAL: NCT01567813
Title: Post-Licensure Observational Study of the Safety of GARDASIL™ in Males
Brief Title: Post-Licensure Study of the Safety of GARDASIL™ in Males (V501-070)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: V501-070; EP08014.070 (Other: Merck)
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Human Papilloma Virus Infection
Keywords: Warts; Papillomavirus infections; DNA virus infections; Virus diseases; Skin diseases, viral; Tumor virus infections; Skin diseases, infectious; Skin diseases
MeSH Terms: conditions — Papillomavirus Infections; Warts; DNA Virus Infections; Virus Diseases; Skin Diseases, Viral; Tumor Virus Infections; Skin Diseases, Infectious; Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Regimen Initiators: Any male health plan member who receives at least one dose of GARDASIL™
- Regimen Completers: Regimen Initiators who complete the 3-dose vaccination regimen within 12 months
- Autoimmune cohort: Regimen Initiators who were members of the health plan during the 12-month period prior to their first dose of GARDASIL™

SUMMARY:
This is a post-licensure safety observation cohort study to describe the general safety of GARDASIL™ (a quadrivalent human papillomavirus vaccine) in males.

ELIGIBILITY:
Inclusion criteria:

* Male vaccinated with at least one dose of GARDASIL™ after the October 2009 FDA date of first licensure of GARDASIL™ for males

Exclusion criteria all cohorts:

* Female
* Male vaccinated prior to the October 2009 FDA date of first licensure of GARDASIL™ for males
* Male who received all doses of GARDASIL™ outside of the health plan

Exclusion criteria, Regimen Completers cohort:

* Male < 9 and > 26 years of age at first dose
* Male not part of health plan at each dose
* 3-dose vaccination regimen given over a period > 12 months
* Less than 28-day interval between first and second dose
* Less than 12 weeks between the second and third dose
* Less than 24 weeks between first and third dose

Exclusion criteria, Autoimmune cohort:

- Male with less than 12 months of health plan membership prior to first dose of GARDASIL™

Ages: 9 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Males who are members of a large geographically diverse US health plan.
Sampling Method: Probability Sample
Enrollment: 114035 (Actual)
Dates: Start 2011-06-23 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of health outcomes resulting in emergency room visits or hospitalizations in 60-day risk periods after each dose of GARDASIL™ compared to post-vaccination self-comparison periods | Within 60 days after each dose

SECONDARY OUTCOMES:
Incidence of health outcomes resulting in emergency room visits or hospitalizations in the 60-day risk period following the first dose of GARDASIL™ compared to post-vaccination self-comparison periods | Within 60 days after the first dose
Incidence of syncope, convulsive syncope, epilepsy, convulsions, head trauma, and allergic reactions on the day of vaccination | Day of vaccination for each dose received (1 day for each dose, up to 3 total days)
Incidence of pre-specified new-onset conditions identified from the hospital, outpatient, and emergency room setting for 6 months after each dose of GARDASIL™ compared to the incidence of these conditions in an un-vaccinated population of males | Within 6 months after each dose

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Amend KL, Turnbull B, Zhou L, Marks MA, Velicer C, Saddier P, Seeger JD. Safety of 4-valent human papillomavirus vaccine in males: a large observational post-marketing study. Hum Vaccin Immunother. 2022 Nov 30;18(5):2073750. doi: 10.1080/21645515.2022.2073750. Epub 2022 Jun 17. PMID 35714277
- [Derived] Seeger JD, Amend KL, Turnbull BR, Zhou L, Marks MA, Velicer C, Saddier P. Incident autoimmune conditions among males receiving quadrivalent human papillomavirus vaccine in the United States. Vaccine. 2023 Mar 10;41(11):1826-1833. doi: 10.1016/j.vaccine.2022.10.050. Epub 2022 Nov 21. PMID 36424257